CLINICAL TRIAL: NCT03208959
Title: A Phase I, Open-Label, Multicenter, Non-Randomized, Dose-Escalation Study to Evaluate the Safety and Tolerability of HTI-1090 in Patients With Advanced Solid Tumors
Brief Title: A Trial of HTI-1090 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTI-1090-101
Record Dates: First submitted 2017-04-26; First posted 2017-07-06 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2019-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose level 1 (Experimental): HTI-1090 tablets will be orally administered on an empty stomach,twice daily, BID i.e., dosing will be 12 hours apart and at approximately the same times each day
  Interventions: Drug: HTI-1090
- Dose level 2 (Experimental): 100% Increment from dose level 1
  Interventions: Drug: HTI-1090
- Dose level 3 (Experimental): 100% Increment from dose level 2
  Interventions: Drug: HTI-1090
- Dose level 4 (Experimental): 100% Increment from dose level 3
  Interventions: Drug: HTI-1090
- Dose level 5 (Experimental): 50% Increment from dose level 4
  Interventions: Drug: HTI-1090

INTERVENTIONS:
Drug: HTI-1090 — IDO/TDO inhibitor
  Other Names: SHR9146

SUMMARY:
IDO1 is expressed in a wide variety of human tumors (eg. bladder, breast, colon, DLBCL, HNSCC, lung, ovarian, uterine, renal…), and contributes to tumoral resistance. HTI-1090 (also referred as SHR9146 in nonclinical study reports) is an orally bioavailable, highly potent, novel small-molecule IDO1/TDO dual inhibitor, with favorable preclinical oral bioavailability and safety profiles.

DETAILED DESCRIPTION:
This is an open-label, dose escalation, phase I, study of HTI-1090 (also known as SHR9146), a small molecule that inhibits both indoleamine 2,3-dioxygenase 1 (IDO1) and tryptophan 2,3-dioxygenase (TDO) - two enzymes that catalyze the oxidation of L-tryptophan (Trp) into kynurenine (Kyn), thereby interrupting the immune escape and the attainment of immunologic tolerance. Dose escalation will use a modified "3+3" design and continue until a MTD or RP2D is identified. This study will also characterize the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of HTI-1090 in subjects with advanced solid tumors.

ELIGIBILITY:
To be eligible to participate in this study, each subject must meet all of the following criteria:

1. Provision of signed fully informed consent prior to any study specific procedures
2. Male or female aged 18 years or older
3. Diagnosed (histologically or cytologically) with solid tumors and documented as advanced or metastatic disease for which there is no known effective anti-tumor treatment (refractory to or relapsed from standard therapies)
4. Subjects may have received one prior IDO, or TDO, or IDO/TDO dual inhibitor therapy; PD-1 or PD-L1 inhibitor; or other therapy that targets T cell co-stimulation or co-inhibition more than 4 weeks prior to the first dose of HTI-1090 (Cycle 1, Day 1)
5. An ECOG Performance Status (PS) of 0 or 1
6. Have a life expectancy ≥ 12 weeks from proposed first dose date
7. Patients must have had no recent major surgery, radiotherapy or chemotherapy over the past 28 days and be fully recover from toxicity before dosing
8. Adequate laboratory parameters during the Screening Period as evidenced by:

   * Absolute neutrophil count ≥ 1.5×109/L (1,500/mm3)
   * Platelets ≥ 100×109/L (100,000/mm3)
   * Hemoglobin (Hgb) ≥ 9.0 g/dL (90 g/L)
   * Subjects may be transfused with red blood cells to improve Hgb levels.
   * Total bilirubin ≤ 1.5×ULN (≤ 2×ULN for subjects with liver metastases)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; for subjects with liver metastases, ALT and AST ≤ 5×ULN
   * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min (measured or calculated by Cockcroft-Gault method)
   * Clinically relevant and treatment resistant abnormalities in potassium, sodium, calcium (corrected for plasma albumin) or magnesium
9. Evidence of post-menopausal status, permanent or surgically sterile, or negative serum pregnancy test for female patients of child-bearing potential. Women will be considered post-menopausal if they are over 50 years old and have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments. Permanent sterilization includes hysterectomy and/or bilateral oophorectomy and/or bilateral salpingectomy but excludes bilateral tubal occlusion. Tubal occlusion is considered a highly effective method of birth control but does not absolutely exclude the possibility of pregnancy. (The term occlusion refers to both occluding and ligating techniques that do not physically remove the oviducts). Women who have undergone tubal occlusion should be managed as if they are of child-bearing potential (e.g., undergo pregnancy testing as required by the study). Females of reproductive potential are required to use reliable contraception
10. Patients must have ability to take and retain oral medication and have no malabsorption problems
11. Willing and able to return to treatment center for follow up, as outlined as protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Adverse events | Cycle 1 (each cycle is 21 days)
  Incidence of AEs
Laboratory results | Cycle 1 (each cycle is 21 days)
  Incidence of laboratory abnormalities
Vital signs | Cycle 1 (each cycle is 21 days)
  Incidence of vital sign abnormalities
Electrocardiogram | Cycle 1 (each cycle is 21 days)
  Incidence of ECG abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Icon Cancer Care Centre, South Brisbane, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No